CLINICAL TRIAL: NCT01182844
Title: Obesity - Inflammation - Metabolic Disease: Effect of Lactobacillus Casei Shirota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanessa Stadlbauer-Koellner, MD (Other)
Responsible Party: Sponsor-Investigator, Vanessa Stadlbauer-Koellner, MD, Associate Professor, Medical University of Graz
Organization: Medical University of Graz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: vs09.2008
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome, probiotic
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care
- Lactobacillus casei Shirota (Experimental): 3 bottles of Yakult(R) light per day
  Interventions: Dietary Supplement: Lactobacillus casei Shirota

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei Shirota — 3 bottles of Yakult(R) light per day
  Other Names: Yakult
  Arms: Lactobacillus casei Shirota

SUMMARY:
Obesity and metabolic syndrome are linked by inflammation. Gut flora seems to play an important role in the development of inflammation and metabolic syndrome in obesity. Modulation of gut flora by probiotics has been shown in animal studies to positively influence inflammation and metabolic disturbances.

Lactobacillus casei Shirota is able to decrease metabolic endotoxemia by altering gut flora composition and gut permeability which leads to an improvement in neutrophil function and insulin resistance in obesity.

The aim of the current study is to investigate the effect of Lactobacillus casei Shirota supplementation over 12 weeks on neutrophil function (phagocytosis, oxidative burst and TLR expression) in patients with metabolic syndrome.

Furthermore the investigators aim to investigate the effect of Lactobacillus casei Shirota supplementation over 12 weeks on glucose tolerance, insulin resistance, inflammation, gut flora composition, gut permeability, and endotoxemia in metabolic syndrome

DETAILED DESCRIPTION:
Obesity and metabolic disorders (type 2 diabetes and insulin resistance) are tightly linked to inflammation. Obesity, a pandemic affecting 30-50% of the adult population, is mediated by a variety of genetic and environmental factors. It is well described that cytokines cause insulin resistance which causes hyperinsulinemia and excessive fat storage in adipose tissue and the liver. However, the triggering factor, linking inflammation to metabolic syndrome has not been fully elucidated yet.

Recently it has been hypothesized that the gut flora is an important factor in this vicious cycle of obesity, metabolic disease and inflammation. Firstly, metabolic activities of the gut microbiota facilitates the extraction of calories from ingested dietary substances and helps to store these calories in host adipose tissue for later use. Second, the gut bacterial flora of obese mice and humans include fewer Bacteroidetes and correspondingly more Firmicutes than that of their lean counterparts, suggesting that differences in caloric extraction of ingested food substances may be due to the composition of the gut microbiota. Furthermore, bacterial lipopolysaccharide derived from the intestinal microbiota may trigger inflammation, linking it to high-fat diet-induced metabolic syndrome. High-fat diet induces insulin resistance and oxidative stress in mice and is associated with increased gut permeability. high fat diet induces a low-grade endotoxemia in mice ("metabolic endotoxemia) and infusing endotoxin causes weight gain and insulin resistance. This has also been shown in humans, where patients with fatty liver had a susceptibility to higher gut permeability, possibly causing increased endotoxin levels.

Endotoxin and Lipopolysaccharide-binding protein (LBP) is elevated in obese patients, patients with type 2 diabetes and patients with liver steatosis. Endotoxin causes a significant increase in proinflammatory cytokine production in adipocytes via a TLR mediated pathway, contribution to the proinflammatory state in obesity. Endotoxin levels correlate with adiponectin and insulin suggesting a pathophysiological link between obesity, inflammation and metabolic disease.

As described above, endotoxin is related to increased inflammation and oxidative stress, causing insulin resistance. Adipocytes have been shown to play a dynamic role in regulation of inflammation by producing cytokines via a Toll-like receptor (TLR)/Nuclear Factor kappa B (NFkB) mediated pathway.But not only adipocytes are in a proinflammatory state - also circulating mononuclear cells have been described to be activated. Clinical evidence suggests immune dysfunction in obesity, since obese patients are more prone to infections after surgery, higher incidence of lower respiratory infection which is also underlined by impairment of cell-mediated immune responses in vivo and in vitro and a reduced intracellular killing by neutrophils.

A similar situation has been recently described in alcoholic cirrhosis and alcoholic hepatitis, which is also a proinflammatory condition with impaired innate immunity, leading to infection. Endotoxin has been described as a key mediator and inadequate activation of neutrophils leading to high oxidative burst and energy depletion of the cells with consecutive impaired phagocytic capacity has been described.

The most effective therapy of obesity - weight loss - leads to significant improvement of mononuclear cell activation. However, there is no data available on the effect of weight loss on gut flora, gut permeability and endotoxin.

Since weight loss is usually very hard to achieve, other therapeutic strategies have been tested. Since gut flora seems to be crucial in the development of the vicious cycle of obesity, inflammation and metabolic disease, several studies tried to modify the composition of gut microbiota. In mice treatment with antibiotics improved glucose tolerance by altering expression of genes involved in inflammation and metabolism. A similar result was found in mice treated with a probiotic that increases the number of Bifidobacterium spp., which leads to improved glucose tolerance, insulin secretion and a decrease in inflammatory tone. Finally treatment of mice with a probiotic decreased hepatic insulin resistance via a C-Jun N-terminal Kinase (JNK) and NFkB pathway, supporting the concept that intestinal bacteria induce endogenous signals that play a pathogenic role in hepatic insulin resistance.

Among the vast amount of bacteria described to alter gut flora and exert positive effects on the host, we have chosen to study Lactobacillus casei Shirota several reasons: Firstly this commercially available preparation delivers a high bacterial number in a relatively small volume and is available as a palatable milk drink. Furthermore Lactobacillus casei Shirota has been proven to survive the passage through the stomach and is present in the lower intestinal tract. It has also been shown that this bacterial strain can increases the amount of Lactobacilli and decreases the number of gram-negative organisms in the bacterial flora. This bacterial strain has been shown to be effective in modulating natural killer cell function and neutrophil function.

We hypothesize that Lactobacillus casei Shirota is able to decrease metabolic endotoxemia by altering gut flora composition and gut permeability which leads to an improvement in neutrophil function and insulin resistance in obesity

Specific Aims:

1. To investigate the effect of Lactobacillus casei Shirota supplementation over 12 weeks on neutrophil function (phagocytosis, oxidative burst and TLR expression) in patients with metabolic syndrome.
2. To investigate the effect of Lactobacillus casei Shirota supplementation over 12 weeks on glucose tolerance, insulin resistance, inflammation, gut flora composition, gut permeability, and endotoxemia in metabolic syndrome

Plan of investigations:

Patients:

30 Patients with metabolic syndrome and increased gut permeability will be randomized to either receive food supplementation with a milk drink containing Lactobacillus casei Shirota (3 bottles a day, 65 ml each, containing Lactobacillus casei Shirota at a concentration of 10^8 colony forming units/ml) for twelve weeks or standard medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Informed consent
* Fasting blood glucose >95mg/dL
* Metabolic syndrome defined by the National Cholesterol Education Program (NCEP) Adult Treatment Panel-III (ATP-III) -ATPIII criteria (3 out of 5)

  * Abdominal obesity (waist circumference >102 in men or >88 in women)
  * Elevated blood pressure (>135/>85) or drug treatment for elevated blood pressure
  * Fasting blood glucose >100mg/dL or previously known type 2 diabetes mellitus,
  * High Density Lipoprotein (HDL) cholesterol <40 mg/dL (men) or <50 mg/dL (women) or drug treatment for low HDL cholesterol
  * Triglycerides >150 mg/dL or drug treatment for elevated for high triglycerides
* HbA1C ≤7.0%

Exclusion Criteria:

* Drug treatment for diabetes mellitus
* Liver cirrhosis (biopsy proven) or elevated transaminases (>2x Upper Limit of Normla (ULN))
* Inflammatory bowel disease (Crohns disease, ulcerative colitis)
* Celiac disease
* Alcohol abuse (more than 40g alcohol per day in the history)
* Clinical evidence of active infection
* Antibiotic treatment within 7 days prior to enrolment
* Use of immunomodulating agents within previous month (steroids etc.)
* Concomitant use of supplements (pre-, pro-, or synbiotics) likely to influence the study
* Any severe illness unrelated to metabolic syndrome
* Malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer-Köllner, MD, Principal Investigator — Dept. of Internal Medicine, Medical University of Graz, Austria; Harald Sourij, MD, Principal Investigator — Dept. of Internal Medicine, Medical University of Graz, Austria
Locations (1):
- Dept. of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Stadlbauer V, Leber B, Lemesch S, Trajanoski S, Bashir M, Horvath A, Tawdrous M, Stojakovic T, Fauler G, Fickert P, Hogenauer C, Klymiuk I, Stiegler P, Lamprecht M, Pieber TR, Tripolt NJ, Sourij H. Lactobacillus casei Shirota Supplementation Does Not Restore Gut Microbiota Composition and Gut Barrier in Metabolic Syndrome: A Randomized Pilot Study. PLoS One. 2015 Oct 28;10(10):e0141399. doi: 10.1371/journal.pone.0141399. eCollection 2015. PMID 26509793
- [Derived] Leber B, Tripolt NJ, Blattl D, Eder M, Wascher TC, Pieber TR, Stauber R, Sourij H, Oettl K, Stadlbauer V. The influence of probiotic supplementation on gut permeability in patients with metabolic syndrome: an open label, randomized pilot study. Eur J Clin Nutr. 2012 Oct;66(10):1110-5. doi: 10.1038/ejcn.2012.103. Epub 2012 Aug 8. PMID 22872030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five subjects were screened for the study between January and August 2010; 30 patients were finally included, whereof 28 finished the study (2 dropped out due to withdrawal of informed consent). Five patients did not fulfill the inclusion criterion of fasting glucose above 100 mg/dl at the day of screening any more.
Period: Overall Study
Arm/Group | Control | Lactobacillus Casei Shirota
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Lactobacillus Casei Shirota | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.9) | 51.5 (11.4) | 53.0 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Neutrophil Phagocytosis From Baseline to 3 Months
Description: The Phagotest® (Orpegen Pharma, Heidelberg, Germany) is used to measure phagocytosis by using Fluorescein isothiocyanate (FITC)-labelled opsonized E. coli bacteria.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of monocytes and granulocytes
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
percentage of monocytes and granulocytes | 0.06 (23.98) | 3.48 (18.83)

2. Primary Outcome: Change of Burst (%) From Baseline to 3 Months
Description: The Phagotest® (Orpegen Pharma, Heidelberg, Germany) is used to measure phagocytosis by using FITC-labelled opsonized E. coli bacteria.
  The Phagoburst® kit (Orpegen Pharma, Heidelberg, Germany) is used to determine the percentage of neutrophils that produce reactive oxidants with or without stimulation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
percent | -8.68 (31.40) | -12.69 (32.96)

3. Secondary Outcome: Change in Indices of Glucose Tolerance and Insulin Resistance
Description: change in indices of glucose tolerance and insulin resistance (frequently sampled in an oral glucose tolerance test) at baseline and after 3 months Homeostasis model assessment (HOMA)- Insulin Resistance (IR): HOMA is calculated by [fasting glucose*fasting insulin/22.5] insulin (U/L), glucose (mmol/l) - higher values indicating more severe insulin resistance Quantitativer Insulin Sensitivitäts-Check Index (QUCIKI): QUICKI is calculated by [1/log (insulin0)+log(glucose0)] insulin (mU/L), glucose (mg/dL) - lower values indicating a improvement of insulin sensitivity Insulin Sensitivity Index (ISI): 0.222-00333*BMI - 0.0000779*Ins120 -0.0004222*age insulin (mU/L) lower values indicating a improvement of insulin sensitivity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: no unit - indices
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
no unit - indices
  HOMA-IR | -0.5 (2.2) | 0.1 (1.9)
  QUICKI | 0 (0.03) | 0 (0.05)
  Insulin sensitivity index (ISI) | 0.004 (0.027) | 0.020 (0.019)

4. Secondary Outcome: Change of Gut Permeability From Baseline to 3 Months
Description: Change of gut permeability (lactulose/mannitol-test) from Baseline to 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
ratio | -0.01 (0.05) | -0.01 (00.06)

5. Secondary Outcome: Change in oxLDL (Oxidative Low Density Lipoprotein) From Baseline to 3 Months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
mU/mL | -55 (197) | -32 (74)

6. Secondary Outcome: Change in Interleukin-6 (IL-6) From Baseline to 3 Months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
pg/mL | 0 [-3.47 to 0.98] | -2.98 [-4.53 to -0.13]

7. Secondary Outcome: Change in Interleukin-10 (IL-10) From Baseline to 3 Months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Control | Lactobacillus Casei Shirota
Number analyzed (Participants) | 15 | 13
pg/mL | 0 [-10.64 to 9.89] | -7.05 [-12.08 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 3 months
Arm/Group | Control | Lactobacillus Casei Shirota
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=15) | Lactobacillus Casei Shirota (N=13)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes